CLINICAL TRIAL: NCT00258843
Title: Clinical Safety Evaluation Study of the Sanofi Pasteur's Inactivated Poliomyelitis Vaccine (IMOVAX Polio™) Administered as a Single Booster Dose at 18 Months of Age in Healthy Chinese Children, and as the First Dose of Primary Vaccination at 2 Months of Age in Healthy Chinese Infants.
Brief Title: Safety of Imovax Polio in Chinese Infants and Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IPV17
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Poliomyelitis
Keywords: IMOVAX;; poliomyelitis
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated

ARMS (2):
- Group 1 (Experimental): Children at 18 months of age
  Interventions: Biological: Inactivated Poliomyelitis vaccine
- Group 2 (Experimental): Infants at 2 months of age
  Interventions: Biological: Inactivated Poliomyelitis vaccine

INTERVENTIONS:
Biological: Inactivated Poliomyelitis vaccine — 0.5 mL, intramuscular (IM)
  Other Names: IMOVAX Polio™ (IPV)
  Arms: Group 1
Biological: Inactivated Poliomyelitis vaccine — 0.5 mL, IM
  Other Names: IMOVAX Polio ™ (IPV)
  Arms: Group 2

SUMMARY:
To describe the tolerance in terms of occurrence of serious adverse reactions and severe adverse reactions (injection site and systemic) within eight days after one dose of IMOVAX Polio™ administered in children and infants.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Aged 18 months (18-20 months) on the day of inclusion
* Group 2: Aged 2 months (56-70 days) on the day of inclusion

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood-derived products received in the past 3 months (for Group 1) or since birth (for Group 2)
* Any vaccination in the 4 weeks preceding the trial vaccination (except BCG and Hepatitis B [Hep B] for Group 2)
* Vaccination planned in the 4 weeks following the trial vaccination
* Group 1: Previous booster vaccination against the poliomyelitis infection with the trial vaccine or with another vaccine.
* Group 2: Previous vaccination against the poliomyelitis infection with the trial vaccine or with another vaccine.
* History of poliomyelitis infection (confirmed either clinically, serologically or microbiologically)
* Clinical or serological evidence of systemic illness including Hepatitis B, C and HIV
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of/current seizures
* Febrile illness (axillary temperature ≥ 37.4°C) or acute illness on the day of inclusion

Ages: 2 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2005-11; Primary Completion 2006-02 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Pingle, China

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com